CLINICAL TRIAL: NCT01988636
Title: Assessment of Safety and Immunogenicity of Intravenous Immunization With Radiation Attenuated Plasmodium Falciparum NF54 Sporozoites (PfSPZ Vaccine) in Healthy African Adults
Brief Title: Study of Safety and Effectiveness of Intravenous Immunization With PfSPZ Vaccine in Healthy African Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); Sanaria Inc. (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 999914010; 14-I-N010
Record Dates: First submitted 2013-11-09; First posted 2013-11-20 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2015-08-20

CONDITIONS: Malaria
Keywords: Randomized; Double Blinded; Mali; Malaria; Transmission
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Group 1 (Experimental): Pilot Safety Group- 135000 PfSPZ + 270000 PfSPZ; staggered at Day 0 and 2 weeks
  Interventions: Biological: PfSPZ Vaccine
- Group 4 (Active Comparator): Group to start at week 4 after Group 1 is deemed safe - 5 immunizations of 270000 PfSPZ at weeks 4, 8, 12, 16 and 24
  Interventions: Biological: PfSPZ Vaccine
- Group 5 (Placebo Comparator): Group to receive placebo at same points as Group 4 - 5 immunizations of normal saline at weeks 4, 8, 12, 16 and 24
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: PfSPZ Vaccine — Aseptic, purified, vialed, cryopreserved, radiation attenuated NF54 p.falciparum sporozoites produced by Sanaria, Inc.
  Arms: Group 1; Group 4
Drug: Placebo — Placebo
  Arms: Group 5

SUMMARY:
Background:

- Malaria is caused by small germs carried by mosquitoes. People can get malaria if an infected mosquito bites them. Malaria destroys red blood cells and reduces oxygen in the blood. Most malaria is mild, but severe malaria kills at least 660,000 people each year. About 75% of these are children in Sub-Saharan Africa, most under age 5. Researchers want to find a safe vaccine that helps prevent malaria.

Objectives:

- To see if a new malaria vaccine is well tolerated and effective.

Eligibility:

- Healthy adults 18 35 years old who are not pregnant and live in Mali.

Design:

* Participants will be screened with medical history, physical exam, and blood test. They will also have an ECG. Soft electrodes will be stuck to the skin. A machine will record the heart s electrical signals.
* Study participation will last about 1 year.
* Participants will be randomly placed in 5 groups. Some will get 2 doses of the PfSPZ vaccine weeks apart; some will get 3 or 5 doses of vaccine; some will get 3 or 5 doses of placebo.
* Doses will be given through a needle in the arm directly into the bloodstream. Then participants must stay at the clinic for 2 hours.
* After each dose, participants will return to the clinic several times for blood tests and physical exam.
* A week before the first dose and 2 weeks after the last, participants will take a full course of anti-malaria drugs.
* If a participant gets malaria during the study, they will take another course of anti-malaria drugs.

DETAILED DESCRIPTION:
For decades it is known that humans can be protected against malaria by repeated immunization with radiation-attenuated sporozoites. Traditionally, those sporozoites are administered by exposing the vaccinee to at least 1000 bites of sporozoite-infected irradiated mosquitoes, an approach that is unsuitable for mass vaccination campaigns. Recently, Sanaria Inc. 1 has developed a process for manufacturing, in compliance with current Good Manufacturing Practices (cGMPs) aseptic, purified, radiation attenuated cryopreserved sporozoites from a wellcharacterized isolate of P. falciparum. This product, which is called PfSPZ Vaccine, can be administered by needle and syringe. Previous studies conducted by the Vaccine Research Center, National Institutes of Health (NIH) and the Navy have established that IV administration of PfSPZ Vaccine can induce sterile protection against controlled human malaria infection (CHMI) with a homologous strain of P. falciparum in up to 100% of malaria na(SqrRoot) ve individuals.

The next logical step is to test the safety and immunogenicity of PfSPZ Vaccine in malaria experienced individuals. As an exploratory objective, this study will collect initial data to find out if the vaccine can protect against naturally occurring infection. Here, we propose a randomized double blind controlled trial to assess the safety and immunogenicity of IV administration of PfSPZ Vaccine in African adults.

Subjects will be recruited from a rural village in Mali. The study will be conducted as collaboration among the Malaria Research and Training Center (MRTC, Mali), the Laboratory of Malaria Immunology and Vaccinology (LMIV) National Institute of Allergy and Infectious Diseases (NIAID), and Sanaria, Inc. Group 1 (n=12), will receive 135,000 PfSPZ Vaccine, followed by 270,000 PfSPZ Vaccine 2 weeks later for safety purposes. An independent Data Safety Monitoring Board (DSMB) will determine whether it is safe to proceed with 270,000 PfSPZ Vaccine.

At Study Week 4, Group 4 (n=50) will receive their first of 5 doses of 270,000 PfSPZ Vaccine given at 4, 8, 12, 16, and 24 weeks, alongside Group 5 (n=50) receiving a similar volume placebo. Safety data will be collected at defined time points after each immunization. From Week 28 until Week 48 all subjects will be monitored for parasitemia detected by slide microscopy every 14 days and by passive case detection.

ELIGIBILITY:
* INCLUSION CRITERIA

The subject must satisfy all the following criteria to be eligible for the study:

1. Signed informed consent form (ICF)
2. Aged 18 to 35 years
3. Long term resident of study site (living there for at least 4 years)
4. Willingness to remain resident in the village and to abstain from travel for prolonged periods during the study
5. Willingness to undergo an HIV test and other tests needed for determining exclusion. (In case of a positive test, the clinician will issue a referral letter to the participant to guide him/her to HIV specialist care for appropriate management and follow up).
6. Willingness to take a curative anti-malarial regimen when prescribed by the investigator
7. Willingness to provide blood for safety data.
8. For females: agreement to use reliable contraception (in the setting where this trial takes place documented depot injection of contraceptives, surgical sterilization ; or an implanted device (all with written evidence provided by an appropriately trained physician) is considered reliable contraception) for the duration of the vaccination phase (i.e., from 1 month prior to first vaccination until 1 month after last vaccination)
9. For females: negative pregnancy test at screening and before each vaccination; women found pregnant will not be given subsequent doses but will be followed up for safety reasons

EXCLUSION CRITERIA

1. Use of antimalarials (other than that prescribed by the investigator) or systemic antibiotics with known antimalarial activity within 30 days prior to the first vaccine dose (e.g. Trimethoprim-Sulfamethoxazole, Doxycycline, Tetracycline, Clindamycin, Erythromycin, Fluoroquinolones, or Azithromycin)
2. Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period
3. Prior receipt of a malaria vaccine candidate
4. Recurrent, severe infections other than malaria, and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
5. Use of immunoglobulins or blood products within 3 months prior to enrolment
6. A history of allergic disease or significant reactions against mosquito bites
7. Known allergies or contraindications against Artemether/Lumefantrine, or

   Atovaquone/Proguanil, such as:
   1. Concurrent medication with Neuroleptics, Antidepressants (i.e., Imipramine, Amitryptilline, Clomipramine and others), Drugs used to treat tuberculosis, including Rifampicin and Rifabutine, Macrolide antibiotics (i.e., Erythromycin, Clarithromycin, Azithromycin, Roxitromycin), Fluoroquinolones (i.e., Ciprofloxacin, Moxifloxacin, Levofloxacin), Antimykotics (i.e., Ketoconazole, Itraconazole), Cimetidine, Class IA and class III antiarrhythmics (i.e., Quinidine, Ajmalin, Disopyramid, Amiodaron, Sotalol), Flecainid, Metoprolol, Cisaprid, Terfenadin, Astemizole, and Metoclopramide
   2. Renal impairment
   3. Symptoms of low potassium, and/or low magnesium
   4. A family history of sudden cardiac death, which in the opinion of the investigator was caused by a pre-existing arrhythmia
   5. Known diagnosis or family history of long QT syndrome
   6. Heart disease (i.e., heart failure, arrhythmias)
8. History of cancer (except basal cell carcinoma)
9. History of serious psychiatric condition that may affect participation in the study
10. If female: currently pregnant, lactating and / or breast-feeding
11. Any other serious chronic illness requiring hospital specialist supervision such as diabetes mellitus type 2.
12. Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 60 g per day
13. Suspected or known injecting drug abuse in the 5 years preceding enrolment
14. Any confirmed or suspected immunosuppressive or immune modulating disorder (i.e., asplenia, lupus, rheumatoid arthritis, vasculitis, sclerodermia, diabetes mellitus)
15. Hematuria, proteinuria, glucosuria as detected by urine dip stick above the levels defined in Appendix F
16. Any clinically significant abnormalities on a 12 lead ECG
17. Seropositive for Hepatitis B surface antigen (HBsAg)
18. Seropositive for Hepatitis C virus (antibodies to HCV)
19. Seropositive for HIV
20. Seropositive for Syphilis
21. Sickle cell trait carriage or sickle cell disease
22. Any clinically significant abnormal finding on biochemistry or hematology blood tests, urinalysis or clinical examination
23. Any other significant disease, disorder or finding which, in the opinion of the investigator, may significantly increase the risk to the subject because of participation in the study, affect the ability of the subject to participate in the study or impair interpretation of the study data.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 296 (Actual)
Dates: Start 2013-10-29; Primary Completion 2015-08-20 (Actual); Study Completion 2015-08-20 (Actual)

PRIMARY OUTCOMES:
Assess the safety of repeated IV immunizations with PfSPZ Vaccine | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Healy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- University of Bamako, Bamako, Mali

REFERENCES:
- [Background] Hoffman SL, Billingsley PF, James E, Richman A, Loyevsky M, Li T, Chakravarty S, Gunasekera A, Chattopadhyay R, Li M, Stafford R, Ahumada A, Epstein JE, Sedegah M, Reyes S, Richie TL, Lyke KE, Edelman R, Laurens MB, Plowe CV, Sim BK. Development of a metabolically active, non-replicating sporozoite vaccine to prevent Plasmodium falciparum malaria. Hum Vaccin. 2010 Jan;6(1):97-106. doi: 10.4161/hv.6.1.10396. Epub 2010 Jan 21. PMID 19946222
- [Background] Seder RA, Chang LJ, Enama ME, Zephir KL, Sarwar UN, Gordon IJ, Holman LA, James ER, Billingsley PF, Gunasekera A, Richman A, Chakravarty S, Manoj A, Velmurugan S, Li M, Ruben AJ, Li T, Eappen AG, Stafford RE, Plummer SH, Hendel CS, Novik L, Costner PJ, Mendoza FH, Saunders JG, Nason MC, Richardson JH, Murphy J, Davidson SA, Richie TL, Sedegah M, Sutamihardja A, Fahle GA, Lyke KE, Laurens MB, Roederer M, Tewari K, Epstein JE, Sim BK, Ledgerwood JE, Graham BS, Hoffman SL; VRC 312 Study Team. Protection against malaria by intravenous immunization with a nonreplicating sporozoite vaccine. Science. 2013 Sep 20;341(6152):1359-65. doi: 10.1126/science.1241800. Epub 2013 Aug 8. PMID 23929949
- [Background] Epstein JE, Tewari K, Lyke KE, Sim BK, Billingsley PF, Laurens MB, Gunasekera A, Chakravarty S, James ER, Sedegah M, Richman A, Velmurugan S, Reyes S, Li M, Tucker K, Ahumada A, Ruben AJ, Li T, Stafford R, Eappen AG, Tamminga C, Bennett JW, Ockenhouse CF, Murphy JR, Komisar J, Thomas N, Loyevsky M, Birkett A, Plowe CV, Loucq C, Edelman R, Richie TL, Seder RA, Hoffman SL. Live attenuated malaria vaccine designed to protect through hepatic CD8(+) T cell immunity. Science. 2011 Oct 28;334(6055):475-80. doi: 10.1126/science.1211548. Epub 2011 Sep 8. PMID 21903775
- [Derived] Sissoko MS, Healy SA, Katile A, Omaswa F, Zaidi I, Gabriel EE, Kamate B, Samake Y, Guindo MA, Dolo A, Niangaly A, Niare K, Zeguime A, Sissoko K, Diallo H, Thera I, Ding K, Fay MP, O'Connell EM, Nutman TB, Wong-Madden S, Murshedkar T, Ruben AJ, Li M, Abebe Y, Manoj A, Gunasekera A, Chakravarty S, Sim BKL, Billingsley PF, James ER, Walther M, Richie TL, Hoffman SL, Doumbo O, Duffy PE. Safety and efficacy of PfSPZ Vaccine against Plasmodium falciparum via direct venous inoculation in healthy malaria-exposed adults in Mali: a randomised, double-blind phase 1 trial. Lancet Infect Dis. 2017 May;17(5):498-509. doi: 10.1016/S1473-3099(17)30104-4. Epub 2017 Feb 16. PMID 28216244